CLINICAL TRIAL: NCT03617172
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Assess The Efficacy and Safety of Misoprostol in The Prevention of Recurrence of Clostridium Difficile Infection in Adults
Brief Title: PROCLAIM -- Misoprostol in the Prevention of Recurrent CDI Prevent Recurrence of Clostridium Difficile Infection With Misoprostol
Acronym: PROCLAIM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ryan S. Doster, MD, Assistant Professor of Medicine, Department of Medicine, Division of Infectious Diseases, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 172163; U01TR002398 (NIH)
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Clostridium Difficile
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Drug (Misoprostol) (Experimental)
  Interventions: Drug: Misoprostol 100Mcg Tab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Misoprostol 100Mcg Tab — Two 100mcg capsules twice per day
  Arms: Study Drug (Misoprostol)
Other: Placebo — Two capsules twice per day
  Arms: Placebo

SUMMARY:
A total of 440 patients meeting enrollment criteria with a primary episode of C. Difficile Infection (CDI) will be enrolled across 3 sites. The total study time period for study procedures followed by clinical monitoring is anticipated to be about 24 months (biomarker assays and other analyses may be completed after the 24 month time period). All participants will receive oral antibiotics for CDI under the care of their physician. After consenting to participate in the study, participants will be randomized to receive either misoprostol (200 mcg po BID) or matching placebo for 14 days. Participants will be monitored for a total time-period of approximately 9 weeks with the goal of monitoring for recurrence of CDI during an 8-week follow-up period from the time that the course of antibiotic treatment is completed. Patients will have blood and stool samples (or rectal swabs if participants are unable to provide a stool sample) collected throughout the study to assess adherence, biomarkers, and to confirm recurrence of CDI (if necessary).

ELIGIBILITY:
Inclusion Criteria

1. Episode of CDI, defined as ALL of the following:

   1. ≥3 unformed (loose or watery) stools with a 24-hour period;
   2. A documented positive C. difficile toxin assay (enzyme immunoassay [EIA] or cell cytotoxicity assay) or NAAT for toxigenic C. difficile from a stool sample collected while the subject was symptomatic; and
   3. No other explanation for diarrhea (e.g. laxatives).
2. At the time of enrollment, on a course of oral antibiotics commonly used for treatment of CDI.
3. Be ≥18 years of age.
4. Be able to provide signed and dated informed consent.
5. Must be able to read and understand English.

Exclusion Criteria

1. Have not recovered from primary episode of CDI at time of enrollment, defined as presence of EITHER of the following:

   1. ≥3 unformed (loose or watery) stools during the 24 hours prior to randomization, OR
   2. Abdominal discomfort (more than mild) present during the 24 hours prior to randomization.
2. Have received, or plans to use, any of the following for treatment of the primary episode of CDI:

   1. Any immunotherapy (e.g., intravenous immunoglobulin, bezlotoxumab).
   2. Any toxin-binding therapy (e.g., cholestyramine [Questran], colestipol [Colestid], or colesevelam [Welchol]).
3. Current or planned treatment with prostanoid therapy.
4. Diarrhea caused by another infection or diarrhea caused by an underlying gastrointestinal disorder.
5. Have any contraindication to oral/enteral therapy (e.g., severe nausa/vomiting or ileus).
6. Have an absolute neutrophil count <500/mm3 [1.0 x 109/L] within 30 days of screening.
7. Require or have an anticipated need for mechanical ventilation or vasopressors for hemodynamic support during the study.
8. Pregnant, nursing, or planning to become pregnant.
9. Inability to understand the requirements of the study, inability to abide by the study restrictions.
10. Have any clinically significant medical or surgical condition that in the investigator's opinion could interfere with the administration of study drug, interpretation of study results, or compromise the safety or well-being of the subject.
11. Known hypersensitivity to misoprostol.
12. Be unwilling or unable to follow study procedures (e.g., study visits, swallow the study drug/placebo, provide stool samples and undergo phlebotomy according to the study schedule, and reliably report information by phone), or not have a caregiver who can ensure that study procedures are followed.
13. If female, be pre-menopausal (cessation of menses less than or equal to 1 year) and not surgically/medically sterile or not following acceptable non-hormonal method of birth control such as abstinence, intrauterine device, or barrier control for at least 1 complete menstrual cycle before the screening visit, or not using estrogen/progestin containing products for at least 2 months before the screening visit through discharge from the study.
14. Unreliable access to telephone service to allow for contact with study personnel.
15. Inability to be seen for routine clinical care either as an outpatient or inpatient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to low enrollment the study was closed early.
Period: Overall Study
Arm/Group | Study Drug (Misoprostol) | Placebo
Started | 3 | 3
Completed | 2 | 3
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug (Misoprostol) | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Recurrence of Clostridium Difficile Infection (CDI).
Description: Number of Participants with clinical recurrence of Clostridium Difficile Infection (CDI) in the 8 week follow-up period.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug (Misoprostol) | Placebo
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

2. Secondary Outcome: Number of Recurrences During the Follow-up Period
Description: Number of recurrences during the follow-up period (for those who have a first recurrence during the follow-up time period)
Time Frame: 8 weeks
Measure: Number; unit: number of events
Arm/Group | Study Drug (Misoprostol) | Placebo
Number analyzed (Participants) | 2 | 3
number of events | 0 | 0

3. Secondary Outcome: Time to Resolution of Diarrhea
Description: Time to resolution of diarrhea (TTROD; for those with recurrence)
Time Frame: 8 weeks
Population: These data were not collected because no participants experienced recurrence.
Arm/Group | Study Drug (Misoprostol) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Randomization - Day 62
Description: An adverse event was any unexpected medical occurrence in any study participant administered an investigational product and may or may not have a causal relationship with treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporarily associated with the use of a medical (investigational) product, whether or not considered related to the medical (investigational) product.
Arm/Group | Study Drug (Misoprostol) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03617172/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT03617172/SAP_001.pdf
  • Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT03617172/ICF_003.pdf